CLINICAL TRIAL: NCT05266573
Title: Effects of a Community Based, Task-Oriented Exercise Program on Community-Dwelling Older Adults With Limited Mobility: A 6-month Longitudinal Cohort Study
Brief Title: Exercise for Adults With Limited Mobility
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Youngstown State University (Other)
Responsible Party: Principal Investigator, Nancy Landgraff, Professor, Youngstown State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 109-2013
Record Dates: First submitted 2022-02-14; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Mobility Limitation; Fall
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise Participants with Limited Mobility (Experimental): The task oriented exercise program consists of 45 to 60 minutes of group exercise sessions with the following components:
  Warm Up: Walking which is progressively increased from 6 to 15 minutes. Dual task activity is introduced as tolerated by the participants. Participants are able to utilize assistive devices and there were additional supports provided.
  Stretching, Strengthening and Balance Activities: Gradual progression of activities and repetitions for 30 minutes that are tailored by the exercise instructor to each participant. Exercises are led by the trainer and performed at the balance bar, in a chair, or in standing. Task oriented activities included items such as: weight shifting, forward/backward/side stepping, squats, forward/backward/side leg raises, toe raises, seated trunk rotations, sit to stand, forward trunk bending, arm rotations, and marching.
  Walk/Obstacle Course: The final 6 to 15 minutes included "challenged walking" through an obstacle course.
  Interventions: Other: Exercise Group

INTERVENTIONS:
Other: Exercise Group — The exercise program is led by an individual who has a background in exercise physiology and is trained by the Physical Therapist. The task oriented exercise program consists of 45 to 60 minutes of group exercise sessions with the following components: warm-up period (dual task activity and walking progressively), stretching/strengthening/balance (gradual progression of activities and repetitions for 30 minutes), and obstacle course (6 to 15 minutes of obstacle course and challenged walking).

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a structured and progressive task-oriented, community based exercise program for older adults who have limitations in mobility and examine whether improvements in mobility and quality of life would be seen following completion at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Limitations in mobility as evidenced by 6 Minute Walk Test score of < 499 meters
* Motivation to participate in an exercise program

Exclusion Criteria:

* unable to follow commands
* unstable cardiac status
* greater than minimal assist for mobility

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-01-08 (Actual); Primary Completion 2017-03-10 (Actual); Study Completion 2017-03-10 (Actual)

PRIMARY OUTCOMES:
Change in 6 Minute Walk Test | Baseline to 6 months
  A submaximal exercise test used to assess aerobic capacity and cardiorespiratory fitness.

SECONDARY OUTCOMES:
Change in Activities Balance Confidence Scale | Baseline to 6 months
  Assesses balance confidence in ambulatory adults and can be used as a predictor for future falls in community dwelling older adults.
Change in Short Form 36 | Baseline to 6 months
  A 36-item survey measuring physical function (PF), role limitations due to physical health problems, role limitations due to emotional problems, bodily pain, general health perceptions, energy/fatigue, social functioning, as well as mental health and emotional well-being.
Change in Gait Speed | Baseline to 6 months
  A measure of the time it takes to travel 10 meters at a pace that is normal for the individual.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Landgraff, PhD, Principal Investigator — Youngstown State University
Locations (1):
- Youngstown State University, Youngstown, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nelson ME, Rejeski WJ, Blair SN, Duncan PW, Judge JO, King AC, Macera CA, Castaneda-Sceppa C. Physical activity and public health in older adults: recommendation from the American College of Sports Medicine and the American Heart Association. Med Sci Sports Exerc. 2007 Aug;39(8):1435-45. doi: 10.1249/mss.0b013e3180616aa2. PMID 17762378
- [Background] Alqahtani BA, Sparto PJ, Whitney SL, Greenspan SL, Perera S, VanSwearingen J, Brach JS. Effect of Community-Based Group Exercise Interventions on Standing Balance and Strength in Independent Living Older Adults. J Geriatr Phys Ther. 2019 Oct/Dec;42(4):E7-E15. doi: 10.1519/JPT.0000000000000221. PMID 31592997
- [Background] Rensink M, Schuurmans M, Lindeman E, Hafsteinsdottir T. Task-oriented training in rehabilitation after stroke: systematic review. J Adv Nurs. 2009 Apr;65(4):737-54. doi: 10.1111/j.1365-2648.2008.04925.x. Epub 2009 Feb 9. PMID 19228241
- [Background] Tisher K, Mann K, VanDyke S, Johansson C, Vallabhajosula S. Functional measures show improvements after a home exercise program following supervised balance training in older adults with elevated fall risk. Physiother Theory Pract. 2019 Apr;35(4):305-317. doi: 10.1080/09593985.2018.1444116. Epub 2018 Mar 5. PMID 29505321
- [Background] Skrastins O, Tsotsos S, Aqeel H, Qiang A, Renton J, Howe JA, Tee A, Moller J, Salbach NM. Fitness coordinators' and fitness instructors' perspectives on implementing a task-oriented community exercise program within a healthcare-recreation partnership for people with balance and mobility limitations: a qualitative study. Disabil Rehabil. 2020 Sep;42(19):2687-2695. doi: 10.1080/09638288.2019.1570357. Epub 2019 Feb 10. PMID 30739500
- [Background] Salbach NM, Howe JA, Brunton K, Salisbury K, Bodiam L. Partnering to increase access to community exercise programs for people with stroke, acquired brain injury, and multiple sclerosis. J Phys Act Health. 2014 May;11(4):838-45. doi: 10.1123/jpah.2012-0183. Epub 2013 May 13. PMID 23676952
- [Background] Salbach NM, Howe JA, Baldry D, Merali S, Munce SEP. Considerations for expanding community exercise programs incorporating a healthcare-recreation partnership for people with balance and mobility limitations: a mixed methods evaluation. BMC Res Notes. 2018 Apr 2;11(1):214. doi: 10.1186/s13104-018-3313-x. PMID 29609662
- [Background] Merali S, Cameron JI, Barclay R, Salbach NM. Characterising community exercise programmes delivered by fitness instructors for people with neurological conditions: a scoping review. Health Soc Care Community. 2016 Nov;24(6):e101-e116. doi: 10.1111/hsc.12282. Epub 2015 Oct 7. PMID 26445890
- [Background] Chompoonimit A, Nualnetr N. The impact of task-oriented client-centered training on individuals with spinal cord injury in the community. Spinal Cord. 2016 Oct;54(10):849-854. doi: 10.1038/sc.2015.237. Epub 2016 Jan 12. PMID 26754477
- [Background] Bird ML, Hill K, Ball M, Williams AD. Effects of resistance- and flexibility-exercise interventions on balance and related measures in older adults. J Aging Phys Act. 2009 Oct;17(4):444-54. doi: 10.1123/japa.17.4.444. PMID 19940323